CLINICAL TRIAL: NCT04730102
Title: Rectal Washout in Transanal Total Mesorectal Excision and Presence of Intraluminal Malignant Cells
Status: Completed | Type: Observational
Sponsor: Slagelse Hospital (Other)
Collaborators: Skane University Hospital (Other); Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: SJ-817; 2019-2567 (Other Grant/Funding Number: Stig & Ragna Gorthons Foundation); ALF Region Skåne (Other Grant/Funding Number: Governmental funding of clinical research within the National Health Services)
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Rectal Cancer
Keywords: Rectal washout; transanal total mesorectal excision; rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing rectal washout in transanal mesorectal excision: Patients undergoing rectal washout in transanal mesorectal excision for rectal cancer.
  Interventions: Procedure: Rectal washout

INTERVENTIONS:
Procedure: Rectal washout — Rectal washout is performed intraoperatively before transection and means irrigation of the rectum following the closure of the rectal lumen below the tumour with a purse string suture. Rectal washout is performed with a total of 500 ml sterile water. Fluid samples are collected after every 100 ml by instilling 50 ml of saline after each washout. A sixth sample is collected from the presacral cavity.

SUMMARY:
The study aims to assess the existence of intraluminal malignant cells and the appropriate fluid volume needed to perform rectal washout during transanal total mesorectal excision (taTME) for rectal cancer.

DETAILED DESCRIPTION:
Twenty patients undergoing taTME for rectal cancer is included. Following the closure of the rectal lumen by a purse string suture, rectal washout is performed with a total of 500 ml sterile water. Fluid samples are collected after every 100 ml by instilling 50 ml of saline after each washout. A sixth sample is collected from the presacral cavity. Each sample is cytologically examined by a pathologist and labelled either malignant or non-malignant.

ELIGIBILITY:
Inclusion Criteria:

* Surgery at Slagelse Hospital for rectal cancer with transanal mesorectal excision
* Consent to participate in the study

Exclusion Criteria:

* No consent to participate
* No surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing transanal mesorectal excision at Slagelse Hospital, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-02-09 (Actual)

PRIMARY OUTCOMES:
Existence of intraluminal malignant cells in fluid samples from rectal washout | Intraoperatively
  Positive/negative cytology

SECONDARY OUTCOMES:
Fluid volume needed to perform rectal washout during transanal total mesorectal excision to eliminate intraluminal malignant cells | Intraoperatively
  Positive/negative cytology

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Buchwald, Principal Investigator — Skåne University Hospital, Malmö, Region Skåne, Sweden
Locations (1):
- Slagelse Hospital, Slagelse, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No